CLINICAL TRIAL: NCT03324776
Title: Initiating Mealtime Ultra-Rapid Acting Insulin (Afrezza) in Uncontrolled Type 2 Diabetes Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Model Clinical Research LLC (Other)
Collaborators: Mannkind Corporation (Industry)
Responsible Party: Principal Investigator, Philip Levin, Senior Director of Clinical Research, Model Clinical Research LLC
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AFR-001
Record Dates: First submitted 2017-10-25; First posted 2017-10-30 (Actual); Results first posted 2024-06-26 (Actual); Last update posted 2024-06-26 (Actual); Status verified 2024-06

CONDITIONS: Type2 Diabetes
Keywords: inhaled insulin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Addition of mealtime Afrezza Inhalation Powder (Other): Patients will be instructed to follow a Weekly Treat-to-Target BG Testing Regimen and make Afrezza dose changes according to an Afrezza Titration Algorithm
  Interventions: Drug: Afrezza Inhalant Product

INTERVENTIONS:
Drug: Afrezza Inhalant Product — Mealtime Ultra-Rapid Acting Insulin
  Other Names: Afrezza Inhaled Insulin

SUMMARY:
To examine the effects of adding prandial Afrezza inhaled insulin to patients with type 2 diabetes who are not controlled after at least 6 months of other diabetes treatments including oral agents, basal insulin, or GLP-1 use.

DETAILED DESCRIPTION:
Clinical inertia in intensifying treatment of type 2 diabetes patients occurs in the range of 70% in numerous real world database assessments. The investigator proposes treating patients with Afrezza who have an index hemoglobin A1c (HbA1c) between 7.5% and 11.5% despite being treated with diabetes medications for at least 6 months. The response to Afrezza will be assessed with Continuous Glucose Monitoring Systems (CGMS) studies and initial and follow-up HbA1c's. The goal is to assess how the investigator can rapidly and safely initiate intensification in this patient population, where extensive delays in HbA1c improvement often occur.

ELIGIBILITY:
Inclusion Criteria:

* Adult type 2 diabetes patients age 18 or older
* HbA1c ≥ 7.5% and ≤ 11.5% after at least 6 months treatment with diabetes medication. Treatment may include oral agents, basal insulin or Glucagon-like peptide-1 (GLP-1) in any combination.
* Patient and provider agree not to add additional diabetes medications during the 14 weeks of the study (unless rescue treatment is indicated).

Exclusion Criteria:

* History of asthma, chronic obstructive pulmonary disease (COPD) or smoking within 6 months
* Forced Expiratory Volume in one second (FEV1) under 70% predicted
* Pregnancy
* Active malignancies and/or life expectancy of < 12 months
* Major surgery planned during study period
* Currently using rapid acting insulins - Novolog, Humalog, Apidra
* Prior use of Afrezza in the last 3 months
* Unwilling to test blood glucose before or after each meal
* Exposure to systemic glucocorticoids within 6 weeks of screening
* Severe hypoglycemia in last 6 months or hypoglycemia unawareness
* Any medical condition which, in the opinion of the investigator, would interfere with ability to understand or respond to the administration of inhaled insulin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2017-10-16 (Actual); Primary Completion 2020-06-10 (Actual); Study Completion 2020-06-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Philip Levin, MD, Principal Investigator — Senior Director of MODEL Clinical Research
Locations (1):
- MODEL Clinical Research, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Addition of Mealtime Afrezza Inhalation Powder
Started | 20
Completed | 20
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Addition of Mealtime Afrezza Inhalation Powder: Adults with Type 2 diabetes on a variety of glucose-lowering regimens instructed to add mealtime Afrezza for 3 months and to follow a weekly treat-to-target BG testing regimen, making Afrezza dose changes according to an Afrezza Titration Algorithm
Arm/Group | Addition of Mealtime Afrezza Inhalation Powder
Number analyzed (Participants) | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.4 (10.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 13
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 7
  White | 11
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 20
Hemoglobin A1c (HbA1c) [Mean (Standard Deviation); unit: percentage of HbA1c] | 9.0 (0.94)
Percent of Time Blood glucose (BG) under 70 mg/dL on Continuous Glucose Monitoring System (CGMS) [Mean (Standard Deviation); unit: percentage of time with glucose <70mg/dL] | 1.1 (2.3)

OUTCOME MEASURES:

1. Primary Outcome: Change in Percentage of HbA1c From Baseline to 3 Months
Description: Change in percentage of HbA1c from baseline to 3 months in uncontrolled type 2 diabetes patients initially having HbA1c of 7.5 or higher and 11.5% or lower
Time Frame: Baseline to 3 months
Measure: Mean (Standard Error); unit: change in percentage of HbA1c
Arm/Group | Addition of Mealtime Afrezza Inhalation Powder
Number analyzed (Participants) | 20
change in percentage of HbA1c | 1.6 (0.247)

2. Secondary Outcome: Percentage of Patients With HbA1c Under 7% at 3 Months
Description: Percentage of patients with uncontrolled type 2 diabetes with HbA1c that is under 7% at 3 months
Time Frame: 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Addition of Mealtime Afrezza Inhalation Powder
Number analyzed (Participants) | 20
Participants | 4

3. Secondary Outcome: Percent of Time With Blood Glucose (BG) Under 70 mg/dL on CGMS
Description: Percent of time with BG under 70 mg/dL on CGMS at 3 months in participants with uncontrolled type 2 diabetes.
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: percent of time with glucose <70mg/dL
Arm/Group | Addition of Mealtime Afrezza Inhalation Powder
Number analyzed (Participants) | 20
percent of time with glucose <70mg/dL | 2.6 (2.5)

ADVERSE EVENTS:
Time Frame: 3.5 months
Description: Adverse Events were collected/reviewed at every visit
Arm/Group | Addition of Mealtime Afrezza Inhalation Powder
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol (2018-02-08): https://cdn.clinicaltrials.gov/large-docs/76/NCT03324776/Prot_000.pdf